CLINICAL TRIAL: NCT07001826
Title: Assessment of the Accuracy of Patient Specific Plates for Correction of Maxillary Cant in Facial Asymmetry: A Prospective Clinical Trial
Brief Title: Assessment of the Accuracy of Patient Specific Plates for Correction of Maxillary Cant in Facial Asymmetry
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdulqader Mohammed Ali Al-hawaagi, PhD Candidate, Department of Oral and Maxillofacial Surgery, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMFS 3-3 -15
Record Dates: First submitted 2025-05-14; First posted 2025-06-03 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Facial Asymmetry
Keywords: High-resolution CT scans; Computer-aided design (CAD); Virtual surgical planning (VSP); Orthognathic surgery; Asymmetrical mandibular deformities; Maxillary cant; LeFort I osteotomy; Bilateral sagittal split osteotomy (BSSO); Patient-specific plates (PSPs); 3D superimposition; Patient satisfaction
MeSH Terms: conditions — Facial Asymmetry; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VSP with Patient-Specific Plates (Experimental): Participants in this arm will undergo orthognathic surgery for correction of maxillary cant using Virtual Surgical Planning (VSP) and custom-designed Patient-Specific Plates (PSPs). The procedure includes preoperative 3D imaging, virtual planning, 3D-printed surgical guides, and personalized fixation plates for precise bone repositioning.
  Interventions: Procedure: Virtual Surgical Planning (VSP) with Patient-Specific Plates (PSPs)

INTERVENTIONS:
Procedure: Virtual Surgical Planning (VSP) with Patient-Specific Plates (PSPs) — Patients will undergo orthognathic surgery using Virtual Surgical Planning (VSP) combined with custom-fabricated Patient-Specific Plates (PSPs). High-resolution CT scans will be used to create 3D models of each patient's craniofacial structure. Surgical plans will be developed using specialized CAD software, and PSPs will be designed and manufactured using 3D printing and milling techniques. During surgery, these custom plates and accompanying cutting guides will be used to accurately reposition the maxilla, ensuring precise correction of maxillary cant. This approach aims to improve surgical accuracy, reduce operating time, and enhance postoperative outcomes.

SUMMARY:
The goal of this clinical trial is to learn how accurate patient-specific plates (PSPs) are for correcting a tilted upper jaw (maxillary cant) in people with facial asymmetry. The main questions it aims to answer are:

* How closely does the actual surgery match the virtual surgical plan?
* How satisfied are participants with how they look after surgery?

Researchers will compare the surgery results using PSPs to the original 3D virtual plan to see how well they match.

Participants will:

* Have a CT scan and 3D virtual surgery planning
* Get custom-made plates designed to fit their upper jaw
* Undergo surgery to correct the tilt of the upper jaw
* Be followed for up to 6 months to check healing and results

DETAILED DESCRIPTION:
This prospective clinical trial aims to evaluate the accuracy and efficacy of patient-specific plates (PSPs) created through virtual surgical planning (VSP) for the correction of maxillary cant in patients with facial asymmetry. Facial asymmetry, particularly in the upper third of the face, often presents with occlusal canting that poses both aesthetic and functional challenges. Traditional orthognathic techniques, such as LeFort I osteotomy with standard fixation hardware, often rely heavily on surgeon experience, potentially compromising consistency and precision.

Virtual Surgical Planning and 3D-Printed PSPs introduce a paradigm shift by enabling surgeons to simulate the osteotomy and repositioning process in a digital environment. This planning facilitates the design and fabrication of custom titanium plates and cutting guides precisely tailored to the patient's skeletal anatomy. This trial investigates whether these individualized devices can achieve closer adherence to the preoperative virtual plan, thus improving surgical accuracy and outcomes.

A sample of eight clinical cases will be included, all diagnosed with maxillary cant and facial asymmetry and meeting defined inclusion/exclusion criteria. The intervention involves a multi-step process:

CT Imaging and Data Acquisition: High-resolution scans of each patient's craniofacial skeleton are obtained in DICOM format.

3D Modeling and Segmentation: Specialized software (Mimics, ProPlan, 3-Matic) is used to segment anatomical structures and perform virtual surgical planning.

Design of PSPs and Surgical Guides: Custom plates and cutting guides are generated based on the planned osteotomy and repositioning.

3D Printing and Manufacturing: Plates are fabricated from titanium using milling techniques, while guides are printed with biocompatible resin.

Surgical Execution: The LeFort I osteotomy, combined with BSSO when indicated, is performed using the guides to ensure precise bone cuts and the PSPs for fixation in the planned position.

The primary outcome is the degree of congruence between preoperative virtual plans and postoperative outcomes, assessed through 3D superimposition of CT images at multiple timepoints (1 week, 1 month, 3 months, and 6 months). Secondary outcomes include aesthetic evaluation and patient satisfaction.

Postoperative care involves standardized antibiotic, analgesic, and steroid regimens, with structured follow-up. Accuracy is quantified in millimeters using reproducible anatomical landmarks. Data will be analyzed using appropriate parametric or nonparametric tests, depending on distribution.

This study addresses a critical gap in the literature by focusing specifically on the role of PSPs in correcting maxillary cant-a feature of asymmetry often overlooked in prior research. The results are expected to contribute evidence-based insights into improving surgical precision, enhancing patient-specific outcomes, and possibly minimizing intraoperative time and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years

Presence of maxillary cant

Presence of facial asymmetry

Exclusion Criteria:

Diagnosis of craniofacial syndrome

History of maxillofacial tumors

History of facial trauma

Presence of cleft lip and/or palate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
To compare pre-operative virtual surgical planning data with post-operative outcomes to measure the correlation between planned and actual surgical results through superimposing of post with planned. | 6 months post-surgery
  performed by superimposing the planned 3D model onto the postoperative 3D model, typically by selecting three or more points to create a plane on the planned model. These same points are then used on the corresponding postoperative model, allowing for an accurate comparison. This method is useful for detecting the accuracy of planning, particularly in assessing pitch and roll movements.
  The accuracy was evaluated using linear measurements (in millimeters), based on specific reproducible points identified on the 3D preoperative casts and compared with the 3D postoperative casts."

SECONDARY OUTCOMES:
To assess the aesthetic outcomes post-treatment, including patient satisfaction | 6 months post-surgery
  Assessment of patient satisfaction using a Likert-scale-based questionnaire evaluating perceived aesthetic and functional improvement.

CONTACTS AND LOCATIONS:
Overall Officials: abdulqadr M al-hawaagi, M.Sc., Principal Investigator — CARIO
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt